CLINICAL TRIAL: NCT06104488
Title: A Multi-Center Phase I Dose Escalation Study of Avutometinib, a RAF/MEK Clamp, in Pediatric Patients With Refractory or Recurrent Solid Tumors Harboring Activating MAPK Pathway Alterations
Brief Title: A Study of Avutometinib for People With Solid Tumor Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 23-129
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Refractory Cancer; CNS Tumors; CNS Tumor, Adult; CNS Tumor, Childhood; MAP Kinase Family Gene Mutation; NF1; Plexiform Neurofibroma; Low-grade Glioma; Optic Pathway Gliomas; Neuroblastoma; Primary Brain Tumor; Solid Tumor; Solid Tumor, Adult; Solid Carcinoma; Central Nervous System Tumor
Keywords: Refractory Cancer; Central nervous system tumor; CNS tumor; Plexiform Neurofibroma; Low-grade Glioma; Optic Pathway Gliomas; Neuroblastoma; Primary Brain Tumor; Solid Tumor; Solid Carcinoma; Avutometinib; Memorial Sloan Kettering Cancer Center; 23-129
MeSH Terms: conditions — Neoplasms; Central Nervous System Neoplasms; Neurofibroma, Plexiform; Neuroblastoma; Brain Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Level -1 (Experimental): If 0 of 3-6 or no more than 1 of 6 evaluable participants experience a DLT, then the dose will be escalated to Dose Level 2 and the same approach will be repeated. If 2 or more DLTs are observed on Dose Level 1 in 2-6 subjects, then further enrollment to Dose Level 1 will stop, the dose will be de-escalated to Dose Level -1 and the same approach will be repeated. The MTD will be the highest dose with <2 DLTs in 6 patients.
  Interventions: Drug: Avutometinib
- Dose Level 1 (Experimental): If 0 of 3-6 or no more than 1 of 6 evaluable participants experience a DLT, then the dose will be escalated to Dose Level 2 and the same approach will be repeated. If 2 or more DLTs are observed on Dose Level 1 in 2-6 subjects, then further enrollment to Dose Level 1 will stop, the dose will be de-escalated to Dose Level -1 and the same approach will be repeated. The MTD will be the highest dose with <2 DLTs in 6 patients.
  Interventions: Drug: Avutometinib
- Dose Level 2 (Experimental): If 0 of 3-6 or no more than 1 of 6 evaluable participants experience a DLT, then the dose will be escalated to Dose Level 2 and the same approach will be repeated. If 2 or more DLTs are observed on Dose Level 1 in 2-6 subjects, then further enrollment to Dose Level 1 will stop, the dose will be de-escalated to Dose Level -1 and the same approach will be repeated. The MTD will be the highest dose with <2 DLTs in 6 patients.
  Interventions: Drug: Avutometinib

INTERVENTIONS:
Drug: Avutometinib — Participants will receive oral avutometinib once daily twice a week, three weeks on/ 1week off, for a period of 28 days per cycle

SUMMARY:
The purpose of this study is to find out whether avutometinib is a safe treatment for advanced or recurrent solid tumor cancers in children and young adults. Researchers will look for the highest dose of avutometinib that is safe and cause few or mild side effects.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible to enroll in this study:

* Age ≥ 3 year and ≤ 30 years at the time of informed consent. *Patients over 18 years of age will be treated at the adult RP2D. The accrual for patients >18 and ≤ 30 years will be limited to no more than 5 patients overall and will not participate in the dose escalation.
* All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.
* Karnofsky ≥ 50% for patients > 16 years of age and Lansky ≥ 50 for patients ≤ 16 years of age.
* Participants must have one of the following:

  1. Histologically confirmed diagnosis of a pediatric tumor including CNS tumors with activating MAP kinase pathway alterations including but not limited to BRAF/ARAF/CRAF fusions or mutations, KRAS/NRAS/HRAS alterations, PTPN11 or SOS1/2 mutations and/or loss of function alterations in NF1. This will be performed at the enrolling institution and central review is not required.

     OR
  2. Participants with a clinical or molecularly confirmed (germline alteration positive) diagnosis of NF1 with symptomatic inoperable plexiform neurofibromas and recurrent/progressive low-grade gliomas are eligible and may enroll without tissue/biopsy confirmation.

OR c) Patients with recurrent optic pathway gliomas are eligible if they have clinical progression (defined as new or worsening neurologic symptoms including visual dysfunction, as defined below):

* Visual worsening, defined as worsening of visual acuity (VA) or visual fields (VF) documented within the past year (by examination or history); OR - Significant visual dysfunction (defined as VA worse than normal for age by 0.6 logMAR [20/80, 6/24, or 2.5/10] or more in one or both eyes).

Molecular testing requirements: Genetic alterations (SNVs or fusions) may be identified through local testing in a Clinical Laboratory Improvement Amendments (CLIA) laboratory in the US or equivalently accredited diagnostic lab outside the United States (US) (CLIA certified) by using molecular assays on any tumor samples (either at initial diagnosis or recurrence). Only the following test modalities are permitted:

* Tissue-based or liquid biopsy NGS or quantitative polymerase chain reaction (qPCR) or RNA based fusion detection (ARCHER or other similar platform).

The reports should be collected for any participants who have completed Next Generation Sequencing (NGS) at any point prior to or during study participation

* Fluorescence in situ hybridization (FISH)
* For subjects enrolled by a liquid biopsy test; blood samples will be required and should be sent prior to enrollment and used for retrospective confirmation in the Sponsor's designated central laboratory (MSKCC).
* Patients must meet the following disease status criteria:
* Solid tumor: Patients must have either measurable disease as measured by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (Version 1.1) or evaluable disease.
* Neuroblastoma subjects are permitted to have evaluable disease only (e.g., bone disease only, evaluable by MIBG or PET).
* Primary Brain Tumors: Patients with primary brain tumors are eligible and can either have measurable disease (defined as at least equal or greater than twice the slice thickness in two perpendicular diameters on MRI) OR evaluable disease (clear MRI evidence of disease that may not be measurable in two perpendicular diameters) OR diffuse leptomeningeal disease OR positive CSF cytology alone.
* Tumor is refractory or recurrent/progressive after standard therapy (at least one prior standard therapy appropriate for tumor type and stage of disease) unless available standard therapies are considered inadequate for the patient.

Exception: NF1 patients with symptomatic and inoperable plexiform neurofibromas that are radiographically progressive or causing significant cosmetic disfigurement or causing significant morbidity are eligible regardless of prior MEK inhibitor exposure

* Patients must have a body surface area (BSA) ≥ 0.67 m2 for enrollment at dose levels 1 and 2) and BSA ≥ 0.83 m2 for patients enrolling at dose level -1.
* Patients must be able to swallow intact capsules.
* Patients may have received prior treatment with a RAF inhibitor (1st or 2nd generation) or MEK inhibitor but only as monotherapy (regardless of prior response to therapy).
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and meet minimum durations (shown below) from prior therapy.

  1. Anti-cancer agents not known to be myelosuppressive: ≥ 7 days
  2. Anti-cancer and cytotoxic agents known to be myelosuppressive: ≥ 14 days
  3. Immunotherapies (including antibodies, interleukins, interferons, etc.): ≥ 21 days
  4. Adoptive cellular therapies (including modified T cells, vaccines, etc.): ≥ 42 days
  5. Autologous stem cell infusion (boost, no conditioning): ≥ 21 days
  6. Autologous stem cell transplantation (with conditioning): ≥ 42 days
  7. Allogeneic bone marrow transplantation: ≥ 84 days
  8. Focal external beam radiation (e.g., limited sites of disease): ≥ 14 days
  9. Substantial external beam radiation (e.g. whole lung or abdomen): ≥ 42 days
  10. Radiopharmaceutical therapy (e.g., radiolabeled antibody or MIBG): ≥ 42 days
* Adequate hepatic function (within 28 days prior to C1D1), defined as:

  1. total bilirubin ≤ 1.5 × upper limit of normal (ULN) for the institution; patients with Gilbert syndrome may enroll if total bilirubin < 3.0 mg/dL (51 μmole/L);
  2. alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN (or < 5x ULN in patients with liver metastases)
  3. Albumin ≥ 3.0 g/dL (451 μmole/L).
* Adequate renal function (within 28 days prior to C1D1) defined a maximum serum creatinine for age and gender defined below. Patients that do not meet the criteria in Table 3 but have a 24 hour Creatinine Clearance or absolute GFR (radioisotope or iothalamate) ≥ 85ml/min are eligible.

Age 1 month to < 6 months: Maximum Serum Creatinine (mg/dL), Male: 0.4; Female: 0.4 Age 6 months to < 1 year: Maximum Serum Creatinine (mg/dL), Male: 0.5; Female: 0.5 Age 1 to < 2 years: Maximum Serum Creatinine (mg/dL), Male: 0.6; Female: 0.6 Age 2 to < 6 years: Maximum Serum Creatinine (mg/dL), Male: 0.8; Female: 0.8 Age 6 to < 10 years: Maximum Serum Creatinine (mg/dL), Male: 1; Female: 1 Age 10 to < 13 years: Maximum Serum Creatinine (mg/dL), Male: 1.2; Female: 1.2 Age 13 to < 16 years: Maximum Serum Creatinine (mg/dL), Male: 1.5; Female: 1.4

≥ 16 years: Maximum Serum Creatinine (mg/dL), Male: 1.7; Female: 1.4 Table 3. The threshold creatinine values in this Table were derived from the Schwartz formula for estimating GFR Schwartz et al. J. Peds, 106:522, 1985) utilizing child length and stature data published by the CDC.

* Adequate hematologic function (within 7 days prior to C1D1), defined as:

  1. platelets ≥100,000/mm3; and
  2. absolute neutrophil count (ANC) ≥ 1000/mm3. Note: Patients may not receive platelet transfusions nor hematopoietic growth factor support, including granulocyte-colony stimulating factor (e.g. filgrastim) and platelet stimulators (e.g. romiplostim) for at least 7 days prior to demonstrating adequate hematologic function.Patients with known malignant bone marrow infiltration are exempt from the above count requirements but should be discussed with sponsor.
* Creatine phosphokinase (CPK) ≤ 2.5 x ULN.
* Adequate recovery from toxicities related to prior treatments to at least Grade 1 by CTCAE v 5.0. Exceptions include alopecia and peripheral neuropathy grade ≤ 2.
* Males or females of reproductive potential must agree to use an effective method of birth control, including a medically accepted barrier or contraceptive method (e.g., male or female condom) for the duration of the study. Abstinence is an acceptable method of birth control until one month after the last dose for female patients and 3 months after the last dose for male pts. Male patients should follow the same direction for sperm donation.

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not eligible to enroll in this study:

* History of rhabdomyolysis.
* Concurrent ocular disorders:

  * Patients with history of glaucoma, history of retinal vein occlusion (RVO), predisposing factors for RVO, including uncontrolled hypertension, uncontrolled diabetes.
  * Patients with history of retinal pathology or evidence of visible retinal pathology that is considered a risk factor for RVO, intraocular pressure > 21 mm Hg as measured by tonometry, or other significant ocular pathology, such as anatomical abnormalities that increase the risk for RVO.
  * Patients with a history of corneal erosion (instability of corneal epithelium), corneal degeneration, active or recurrent keratitis, and other forms of serious ocular surface inflammatory conditions.
* Patients with a history of hypersensitivity to any of the inactive ingredients (hydroxypropylmethylcellulose, mannitol, magnesium stearate) of the investigational product.
* Ongoing active diarrhea requiring medication (e.g., loperamide, bile acid sequestrant such as cholestyramine) within 7 days.
* Clinically significant cardiac disease or risk factors at screening including any of the following:

  1. Any history of congestive heart failure
  2. Left ventricular ejection fraction (LVEF) < 50% or below the institutional standard lower limit, whichever is higher, as determined by multiple gated acquisition (MUGA) scan or Trans-thoracic echocardiography (TTE)
  3. QTc > 470 msec regardless of sex (using Bazett formula) on screening ECG (using triplicate ECGs), history of Torsades de Pointes, or a history of congenital long QT syndrome.
* Known hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection that is active and/or requires therapy.
* Exposure to strong CYP3A4 inhibitors and inducers within 14 days prior to the first dose and during the course of therapy (see appendix A).

  * Known strong and moderate inducers or inhibitors of CYP3A4/5, including enzyme-inducing anti-convulsant drugs (EIACDs), grapefruit, echinacea, grapefruit hybrids, pummelos, starfruit, and Seville oranges.
  * Substrates of CYP3A4/5 with a narrow therapeutic index.
  * Herbal preparations/medications (except for vitamins) including, but not limited to:
  * St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone
  * (DHEA), yohimbe, saw palmetto, black cohosh and ginseng.
* Pregnant or breastfeeding women will not be entered on this study because there is yet no available information regarding human fetal or teratogenic toxicities.

Ages: 3 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2029-10-20 (Estimated); Study Completion 2029-10-20 (Estimated)

PRIMARY OUTCOMES:
Safety of avutometinib | up to 12 months
  The primary objective is to assess the safety of avutometinib in the pediatric population. CTCAE Version 5 will be utilized for toxicity evaluation. Adverse Events should be recorded from treatment start through 30 days after the last dose of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Sameer Farouk Sait, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Children's Healthcare of Atlanta (Data Collection Only), Atlanta, Georgia
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org